CLINICAL TRIAL: NCT04137159
Title: An Exercise Intervention to Educe Neuropathic Pain and Brain Inflammation After Spinal Cord Injury
Brief Title: An Exercise Intervention to Reduce Neuropathic Pain and Brain Inflammation After Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Nils Clas Linnman, Assistant Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019P003113
Record Dates: First submitted 2019-10-18; First posted 2019-10-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized cross-over wait-list controlled
Who Masked: Outcomes Assessor
Masking Description: Study statistician is masked to intervention type
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FES rowing (Experimental): Exercise training sessions will be performed 3 times per week for 12 weeks. The initial training sessions will include 6 sets of FES-rowing for 5 min at 60% of VO2 peak with a work-to-rest ratio of 2:1. Participants unable to row continuously for 5 min will row for 2-4 min with 30-second breaks incorporated until they achieve sets totaling 30 min. The goal is for each volunteer to achieve an exercise intensity of 70-85% maintained for a continuous 30-40 min performed 3 times each week.
  Interventions: Other: Functional Electrical Stimulation rowing exercise
- Wait list (No Intervention): During the 12-week treatment as usual program, subjects will not participate in FES-rowing.

INTERVENTIONS:
Other: Functional Electrical Stimulation rowing exercise — Full-body aerobic exercise
  Arms: FES rowing

SUMMARY:
Spinal Cord Injury (SCI) leads to alterations in brain structure and function by spinal nerve damage, secondary inflammatory responses, and by the consequences of living with paralysis and neuropathic pain. Physical inactivity due to lower body paralysis rapidly leads to loss of muscle, and risk of heart disease. The leading cause of death after a spinal cord injury is cardiovascular disease, and just a year after injury, those with SCI have a peak exercise capacity half that of the unfit general population.

The good news is that aerobic exercise reduces the risk of chronic metabolic and cardiorespiratory diseases, reduces inflammation and pain, and increases mood and quality of life. Exercise can also reduce brain inflammation, enhance endogenous analgesia, and increases the size of the hippocampus.

The issue is that muscle paralysis in SCI restricts the ability to achieve the levels of exercise that is necessary for broad analgesic, anti-inflammatory and neuroprotective benefits. Arm exercise can have some effects on heart and lung capacity, but the small muscle mass is insufficient to produce more than modest aerobic work. With functional electrical stimulation (FES), leg muscles that are paralyzed can be made to contract, thereby allowing more of the body to be exercised. The full rowing stroke is produced by both the (stimulated) legs and arms, increasing the active muscle mass and resulting in an aerobic work-out that is intensive enough to improve heart, lung, and - maybe - brain function.

In this clinical trial of sub-acute spinal cord injured subjects, the investigators will study how 12 weeks of FES-RT, in comparisons to 12 weeks of wait-list, changes pain, brain structure, endogenous opioid function and brain inflammation.

The investigators will measure changes using positron emission tomography and magnetic resonance imaging. The investigators hypothesize a decrease in pain interference, an increase in hippocampal volume, increased endogenous opioid transmission in the periaqueductal gray, and decreased hippocampus neuroinflammation.

DETAILED DESCRIPTION:
This clinical trial will utilize a randomized, controlled, crossover design. Participants will be randomized to (A) 12 weeks of FES-RT followed by 12 weeks of treatment as usual or (B) 12 weeks of treatment as usual followed by 12 weeks of FES-RT.

Randomization will be computer generated and the study statistician will keep the key to appropriately conceal allocation of treatment until after obtaining baseline measures.

Exercise Intervention:

FES-RT occurs in two distinct steps - an initial strength training step, followed by FES-RT. Those with SCI can require at least two weeks and up to six weeks of strength-training. For the strength training, electrodes are placed over motor points of the quadriceps and hamstrings and intensity of the stimulus is set at the level producing full knee flexion-extension. Training is performed until subjects can complete a flexion extension protocol for 30 min without rest. During this time, the first set of PET-MR data will be obtained.

Subsequently, the FES-RT commences.

Measurements / Assessments Exercise Capacity: Volunteers will perform an incremental exercise test of FES- or arms-only rowing to determine maximal oxygen uptake on a day normally scheduled for regular exercise training. Exercise capacity and aerobic power will be determined from on-line computer-assisted open circuit spirometry. Subjects will row with increasing resistance every 2 min until volitional fatigue. To ensure attainment of maximal exercise capacity, at least 3 of these criteria will be met: 1) O2 consumption plateaus despite increasing workload, 2) respiratory exchange ratio >1.10 at end exercise, 3) age-predicted maximal heart rate is achieved, and 4) perceived exertion is rated at least 16 on the Borg scale of 6-20.

Exercise Volume: The progression of the exercise stimulus across the training program will be assessed from duration, frequency, and intensity derived from heart rate monitored during each exercise bout (i.e., Training Impulses or TRIMPs) as well as the product of average wattage and total duration for each week. TRIMPs are routinely used to quantify the exercise load and is specific to the cardiopulmonary system. The investigators will also calculate exercise load or work as the product of the weekly average of wattage and weekly total of exercise time.

PET-MR imaging

Neuroimaging metrics will be obtained at baseline, after 12 weeks and after 24 weeks. MR-PET scanning will be performed at 3 Tesla, using a Siemens whole-body MRI, whole-body PET camera (Biograph MMR). MRI data will be acquired simultaneously to the PET data.

In response to injury, microglia migrate to the site of injury, and express multiple cell surface proteins, including the translocator protein (18kDa) (TSPO). This conditional expression makes TSPO a prime target for PET imaging (127). There are multiple candidate PET tracers for glial activity , whereof 11C-PBR28 is a sensitive, second generation, high affinity TSPO radioligand suitable for imaging of microglial and astrocytic activation in neuroinflammation in humans. For glial imaging, 11C-PBR28 will be injected intravenously with a slow bolus over a 30s period (130). Dynamic data will be collected over the brain for 90 minutes in list mode, and framed post-collection. The dose will be up to 15mCi, which is equivalent to ~3.7 mSv.

For opioid imaging, 11C-diprenorphine will be injected intravenously, Dynamic data will be collected over the brain for 90 minutes in list mode, and framed post-collection. The dose will be up to 12mCi, which is equivalent to ~2.5 mSv.

For both scans, MR-based attenuation correction maps are created based on the MPRAGE data. For glial imaging, standardized uptake values (SUV), normalized to whole brain PBR28 ligand uptake, will be used. For 11CDiprenorphine, kinetic modeling is carried our using subject specific bilateral occipital cortices as the reference tissues. Nondisplaceable binding potential maps (BPND), representing the relative amount of specifically bound radioligand to that of non-displaceable radioligand, are calculated from the 90 min of dynamic PET data using a simplified reference tissue model with the occipital cortex used as the reference tissue.

A high resolution structural volume will be collected for the purposes of longitudinal structural analyses. All longitudinal data analyses will be done in native space as repeated measurements, thereby avoiding spatial normalization errors typically associated with cohort studies.

A battery of pain, quality of life and psychological well-being questionnaires to the participants on four occasions: immediately after enrollment, at the start of the 12 week wait-list or FES-RT period, at the end of the first arm, and at the end of the cross-over arm (24 weeks).

Conditioned pain modulation: Conditioned pain modulation (CPM) is a psychophysically-based laboratory method to reliably ) evaluate the individual capabilities to inhibit pain in humans. Briefly, CPM is based on the "pain inhibits pain" phenomenon when Stimulus A (test-pain) given together with Stimulus B (conditioning pain) is perceived less painful than when Stimulus A was given alone. Although the literature is not entirely consistent, CPM can be reduced with naltrexone, suggesting at least partial dependence of inhibition on endogenous opioids. CPM will be determined at baseline, 12 weeks and 24 weeks, with the hypothesis that FES-RT will lead to increased CPM.

ELIGIBILITY:
Inclusion Criteria:

* SCI at or below neurological level C5 with American Spinal Injury Association grade A, B or C, within 3-24 months after injury.

Exclusion Criteria:

* pregnancy
* breast feeding
* contraindications to MRI
* contraindications to PET current or past history of:
* major medical illness
* major neurological illness other than SCI
* major psychiatric illness
* diabetes
* major kidney or liver problems
* use of tobacco
* use of recreational drugs
* an abnormal physical exam (e.g., heart murmurs or peripheral edema).
* unresponsive to FES stimulation
* heart disease
* physical limitations to FES-RT success
* blood pressure>140/90 mmHg
* significant arrhythmias
* cancer
* epilepsy
* current use of cardioactive medications
* current grade 2 or greater pressure injuries at relevant contact sites
* peripheral nerve compressions or rotator cuff tears that limit the ability to row
* history of bleeding disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Change in PROMIS Pain Interference questionnaire | Change between baseline and after 12 week FES intervention, and after 12 week wait list
  The Patient-Reported Outcomes Measurement Information System (PROMIS(r)) Pain Interference instrument measure the self-reported consequences of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Pain Interference also incorporates items probing sleep and enjoyment in life.
  The scale ranges from 6 to 30, with 30 being the highest pain interference.
Change in Hippocampal volume | Change between baseline and after 12 week FES intervention, and after 12 week wait list
  MRI derived measurement of hippocampus volume
Change in Hippocampus glial activation | Change between baseline and after 12 week FES intervention, and after 12 week wait list
  11C-PBR28 SUV uptake in the hippocampus
Change PAG opioid binding potential | Change between baseline and after 12 week FES intervention, and after 12 week wait list
  Non-displaceable opioid binding potential of the periaqueductal gray

CONTACTS AND LOCATIONS:
Overall Officials: Nils C Linnman, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No HIPAA protects data will be shared. Neuroimaging data may be shared.